CLINICAL TRIAL: NCT05108337
Title: Ultrasound Guided Superficial Cervical Plexus Block for Chronic Pain After Craniotomy Via Suboccipital Retrosigmoid Approach: A Randomized Controlled Trial
Brief Title: Superficial Cervical Plexus Block for Postoperative Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, MD,PhD, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-10-16
Record Dates: First submitted 2021-10-21; First posted 2021-11-04 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Neurosurgery
Keywords: Cervical Plexus Block; Chronic pain; Neurosurgery
MeSH Terms: conditions — Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scpb group (Experimental): Superficial cervical plexus block group
  Interventions: Procedure: Superficial cervical plexus block
- Control group (Sham Comparator): Saline group
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: Superficial cervical plexus block — Ultrasound guidance will be used to determine the location of superficial cervical plexus nerve. The puncture will also be performed by ultrasound guidance, covered with opaque infusion dressing but performed with infusion of 10 ml 0.5% ropinacaine.
  Arms: Scpb group
Other: Control group — Ultrasound guidance will be used to determine the location of superficial cervical plexus nerve. The puncture will also be performed by ultrasound guidance, covered with opaque infusion dressing but performed with infusion of 10 ml normal saline.
  Arms: Control group

SUMMARY:
The incidence of postoperative chronic pain after craniotomy is high. Postoperative chronic pain seriously affects patient's quality of life. Compound local scalp nerve block is a good choice for analgesia after craniotomy. However, the scalp nerve block commonly cannot cover the area of suboccipital retrosigmoid approach craniotomy, leading to incomplete block. Superficial cervical plexus block (SCPB) is theoretically promising to solve the analgesia requirements of such surgical approach. At the same time, ultrasound guidance can not only accurately locate, ensure the effect of block and avoid accidental injury during puncture. The purpose of this study is to explore whether ultrasound-guided superficial cervical plexus block can safely and effectively reduce the incidence of chronic pain after craniotomy via suboccipital retrosigmoid approach.

ELIGIBILITY:
Inclusion Criteria:

1. Elective suboccipital retrosigmoid approach approach craniotomy;
2. Age between 18 and 65 years;
3. American Society of Anesthesiologists (ASA) physical status I-III.

Exclusion Criteria:

1. The patients or legal clients refuse to provide informed consent;
2. Local infection;
3. Preoperative impairment of consciousness and cognitive function;
4. Uncontrolled hypertension;
5. Inability to communicate;
6. Allergies to experimental drugs;
7. History of drug abuse;
8. History of chronic headache;
9. Aphasia and hearing impairment;
10. Patients undergoing second craniotomy;
11. Body mass index < 18.5 kg/m2 or > 35.0 kg/m2;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Chronic pain assessment | at 3 months after surgery.
  Follow-up visit will be conducted by telephone at 3 months after surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality